CLINICAL TRIAL: NCT00683267
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate Efficacy, Safety, Tolerability, and Pharmacokinetics of a Single Intraoperative Localized Instillation of 4975 in Patients Undergoing Primary Unilateral Total Hip Arthroplasty
Brief Title: Efficacy and Safety Study of 4975 in Patients Undergoing Total Hip Replacement
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment of patients has halted prematurely and will not resume. No future patients will be enrolled or treated.
Sponsor: Anesiva, Inc. (Industry)
Responsible Party: Shaun Comfort, MD, Anesiva, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114-03P
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2009-05-04 (Estimated); Status verified 2009-05

CONDITIONS: Arthroplasty
Keywords: THA, Total hip arthroplasty, total hip replacement
MeSH Terms: interventions — ALGRX-4975

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Study treatment, 4975, is instilled directly into surgical site
  Interventions: Drug: 4975, highly purified capsaicin
- 2 (Placebo Comparator): Placebo is instilled directly into surgical site
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 4975, highly purified capsaicin — One dose administered by direct instillation into the surgical site
  Other Names: 4975, Adlea
  Arms: 1
Drug: Placebo — One dose administered by direct instillation into the surgical site
  Arms: 2

SUMMARY:
Evaluate the efficacy, safety and tolerability of a single intraoperative dose of 4975 in patients undergoing total hip replacement

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of a single intraoperative dose of 4975 in patients undergoing primary unilateral total hip arthroplasty

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female aged 18 to 85 years with an American Society of Anesthesiologists (ASA) status of I, II, III
* Planning to undergo unilateral THA
* In good health and capable of undergoing THA with spinal block and sedation anesthesia
* No additional planned surgeries during the course of the trial
* Willing and able to complete the study procedures and pain scales and to communicate meaningfully in English

Key Exclusion Criteria:

* A body mass index greater than 40
* Known bleeding disorder or is taking agents affecting coagulation preoperatively
* A medical condition that could adversely impact the patient's participation, safety, or conduct of the study
* Diabetes mellitus with a known HbA1C>9.5 or a history of prolonged uncontrolled diabetes
* Previous hip arthroplasty of the same hip
* Participated in another clinical trial within 30 days of the planned hip surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2007-09; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) measures of pain at prespecified times | Primary endpoint is 2 days (4-48 hours)

SECONDARY OUTCOMES:
Other efficacy endpoints, safety and tolerability of 4975 | 42 Days

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Comfort, MD, MBA, Study Director — Anesiva, Inc.; William Houghton, MD, Study Director — Anesiva, Inc.
Locations (10):
- United States (10):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Lotus Clinical Research, Inc., Arcadia, California
  - Glendale Adventist Medical Center, Glendale, California
  - Webster Orthopaedic Medical Group, Oakland, California
  - University of California at San Francisco - Mt. Zion, San Francisco, California
  - Coastal Medical Research, Inc., Port Orange, Florida
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Sewickley Valley Hospial, Sewickley, Pennsylvania
  - Covenant Medical Center, Lubbock, Texas

REFERENCES:
- See also: Anesiva Home page — http://www.anesiva.com/wt/page/pipeline
- See also: ADLEA Product Information — http://www.anesiva.com/wt/page/adlea